CLINICAL TRIAL: NCT06550453
Title: Safety and Efficacy of Pembrolizumab in Combination with Bevacizumab + CapeOX in the Neoadjuvant Treatment of RAS-mutated, BRAF Wild-type, Microsatellite-stabilized, Locally Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: yangjianjun (Other)
Responsible Party: Sponsor-Investigator, yangjianjun, Professor in Xijing Hospital, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20232402
Record Dates: First submitted 2024-08-02; First posted 2024-08-13 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-08

CONDITIONS: Locally Advanced Colorectal Cancer
Keywords: Locally advanced colorectal cancer (LACRC); pembrolizumab; microsatellite-stabilized; CapeOX neoadjuvant
MeSH Terms: interventions — Bevacizumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pembrolizumab + bevacizumab and CapeOX (bevacizumab + oxaliplatin + capecitabine) (Experimental): all enrolled patients received a combination of chemotherapy and immunotherapy, as outlined below:
  Pembrolizumab:
  Day 1：Pembrolizumab injection 200mg was administered once and repeated every 21 days, expected to last 2-4 cycles. Two vials (200 mg) of pembrolizumab injection should be diluted into 100-200 mL of saline, and the infusion time should be more than 30 minutes.
  Chemotherapy (CapeOX regimen):
  Day 2: Bevacizumab (7.5 mg/kg) + Oxaliplatin (135 mg/m2) + Capecitabine (1 g/m2, did, d1-d14). Treatment repeated every 3 weeks (q3w) until disease progression or intolerable toxicity.
  Interventions: Drug: Pabolizumab+ bevacizumab and CapeOX (bevacizumab + oxaliplatin + capecitabine)

INTERVENTIONS:
Drug: Pabolizumab+ bevacizumab and CapeOX (bevacizumab + oxaliplatin + capecitabine) — Pabolizumab is an lgG4 subclass monoclonal antibody humanized against PD-l molecules thatblocks the immune escape mechanism of cancer cells by inhibiting the PD-l receptor oflymphocytes, thereby allowing the immune system to destroy them.
  In the single-arm study, all enrolled patients received a combination of chemotherapy and immunotherapy, as outlined below:
  Pembrolizumab:
  Day 1：Pembrolizumab injection 200mg was administered once and repeated every 21 days, expected to last 2-4 cycles. Two vials (200 mg) of pembrolizumab injection should be diluted into 100-200 mL of saline, and the infusion time should be more than 30 minutes.
  Chemotherapy (CapeOX regimen):
  Day 2: Bevacizumab (7.5 mg/kg) + Oxaliplatin (135 mg/m2) + Capecitabine (1 g/m2, did, d1-d14). Treatment repeated every 3 weeks (q3w) until disease progression or intolerable toxicity.

SUMMARY:
To explore the efficacy and safety of pembrolizumab in combination with bevacizumab and CapeOX neoadjuvant therapy for the treatment of RAS-mutated, BRAF wild-type, microsatellite-stabilized, locally advanced colorectal cancer.

Methods and analysis: A prospective, open-label, single-arm, phase 2 clinical study protocol will enroll a total of 20 patients. The study is designed as a Simon II Optimal study involving 20 locally advanced rectal cancer (LACRC) patients. Initially, 9 patients will be recruited in the Simon I phase, and if more than 1 patient achieves a pathological complete response (pCR), the study will proceed to the II phase. Recruit up to 20 patients in Phase II, and if more than 4 patients achieve pCR, the trial will be considered successful. All enrolled patients will receive 2-4 cycles of neoadjuvant therapy with pembrolizumab + bevacizumab and CapeOX (bevacizumab + oxaliplatin + capecitabine). The primary efficacy endpoint is the pathological complete response (pCR) of the cancer following neoadjuvant therapy. Secondary efficacy endpoints include major pathological response (MPR), objective response rate (ORR), and assessment of adverse events (AEs).

Ethics: Ethics approval has been obtained from the Ethics Committee at the First Affliated Hospital (Xijing Hospital)(KY20232402-F-1)

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years;
* Confirmed RAS mutation and BRAF wild-type in LACRC by pathological histology or genetic sequencing.;
* ECOG Performance Status (PS) score of 0 or 1;
* Previously untreated;
* Microsatellite-stable status;
* Hematological parameters within normal limits: White blood cell count ≥4×10^9/L; Absolute neutrophil count ≥1.5×10^9/L; Platelets ≥100×10^9/L. Hemoglobin ≥90g/L;
* Normal renal function: Serum creatinine ≤1.5× upper limit of normal (ULN) or creatinine clearance (CrCl) >60 mL/min (calculated using Cockcroft-Gault formula): Female CrCl = (140 - age) × weight (kg) × 0.85 / (72 × Scr mg/dl)；Male CrCl = (140 - age) × weight (kg) × 1.00 / (72 × Scr mg/dl);
* Normal liver function: Serum total bilirubin ≤1.5× ULN; Aspartate aminotransferase (AST) ≤2.5× ULN; Alanine aminotransferase (ALT) ≤2.5× ULN;
* Female patients must have a negative pregnancy test before the study initiation (not applicable to bilateral oophorectomy and/or hysterectomy patients or postmenopausal patients);
* Signed written informed consent form.

Exclusion criteria:

* Receiving anti-tumor therapy prior to enrollment, including but not limited to PD-1 inhibitors, CTLA-4 antibodies, EGFR monoclonal antibodies, EGFR-TKI, and anti-angiogenic drugs;
* History of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome-associated vascular thrombosis, Wegener's granulomatosis, desiccation syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. (Note: Vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune disease, psoriasis not requiring systemic therapy, or patients not expected to have a relapse without external triggers may be allowed to enroll);
* Enrolled in another interventional clinical trial within 30 days prior to screening;
* History of other malignancies (except cured basal cell carcinoma of the skin);
* Presence of severe, poorly controlled co-morbidities such as heart failure, diabetes mellitus, hypertension, hepatic failure, renal failure, thyroid disease, psychiatric disorders, etc;
* Known HIV infection or active viral hepatitis or tuberculosis;
* Major surgery or planned surgery within 30 days prior to the first dose of the investigational drug;
* Hypersensitivity to the drugs used in the trial or their components;
* Pregnancy (confirmed by blood or urine HCG test) or breastfeeding women, or subjects of childbearing potential unwilling or unable to use effective contraception until at least 6 months after the last trial treatment;
* Deemed inappropriate for participation in the study by the investigator.
* Unwilling or unable to participate in the study or sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | 12 months
  Pathological complete reand the postoperative pathological findings were statistically completse rate (pCR rate): The pathological status of the primary site was determined in the surgical patient Proportion of patients with complete response:

SECONDARY OUTCOMES:
Objective response rate (ORR) in the neoadjuvant phase | 36 months
  Obiective response rate (ORR) at the neadjuvant stage: proportion of subjects who achieved partiaand complete response on radiographic assessment (RECIST v1.l) after the end of neoadjuvanttherapy;
Major pathological response rate (MPR) | 36 months
  Major pathological response rate (MPR rate): The pathological status of the primary site wadetermined in the patients undergoing surgery, and the proportion of patients with residuatumor cells <10% by pathological detection in postoperative specimens was counted
Adverse event rate (AE) | 36 months
  Safety: all adverse events, serious adverse events;

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affliated Hospital (Xijing Hospital),the First Affiliated Hospital of Air Force Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided